CLINICAL TRIAL: NCT00593242
Title: Autologous Cord Blood Cells for Hypoxic Ischemic Encephalopathy Study 1. Phase I Study of Feasibility and Safety.
Brief Title: Cord Blood for Neonatal Hypoxic-ischemic Encephalopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Cotten (Other)
Responsible Party: Sponsor-Investigator, Michael Cotten, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000412; Duke NPRI01
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Hypoxic Ischemic Encephalopathy
Keywords: hypoxic-ischemic encephalopathy; autologous cord blood cells; newborn infants
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- infusions (Experimental): infants who arrive at the study site within the first 14 postnatal days and had a history of moderate to severe hypoxic ischemic encephalopathy, and have cells available for infusion that pass Carolinas Cord Blood Bank Quality checks Outcomes will be measured at 22-26 months fby neurodevelopment assessment
  Interventions: Biological: infusion of autologous cord blood
- historical control (Other): Infants who had moderate to severe hypoxic ischemic encephalopathy in the neonatal period but did not receive autologous cord blood cells.
  Interventions: Other: Neurodevelopmental outcomes

INTERVENTIONS:
Biological: infusion of autologous cord blood — infants who meet study enrollment criteria for history of moderate to severe hypoxic ischemic encephalopathy in the neonatal period will receive up to 4 infusions of their own volume reduced cord blood cells. The number of doses will be determined by the amount of available cord blood cells. The dose for each infusion is 5x10e7 cells/kg
  Arms: infusions
Other: Neurodevelopmental outcomes — historical controls, no experimental intervention, standard therapies of hypoxic ischemic encephalopathy in the newborn period with autologous cord blood
  Arms: historical control

SUMMARY:
This is a pilot study to test feasibility of collection, preparation and infusion of a baby's own (autologous)umbilical cord blood in the first 14 days after birth if the baby is born with signs of brain injury.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the safety and feasibility of infusions of autologous (the patient's own)umbilical cord blood cells in term gestation newborn infants with hypoxic-ischemic encephalopathy. For this study, infants who have signs of moderate to severe encephalopathy at birth whose mothers have previously consented to providing cord blood cells for the Carolinas Cord Blood Bank or other public or private bank that uses accepted standards for collection and handling of cells, or provided verbal consent for cord blood collection for the possibility of their baby's participation in this trial, can receive their own cord blood cells if an adequate number of cells that meet Carolinas Cord Blood Bank Quality standards are available in the first 14 postnatal days. Study activities also include serial blood draws concurrent with clinically indicated blood draws with a total volume of no more than 5 milliliters (1 teaspoon) from all study related tests. Babies will be followed for neurodevelopmental outcome at 4 - 6 and 9 - 12 months at Duke's Special Infant Care Clinic. MRI's will be obtained per clinical routine and results will be analyzed and described in study reports.

ELIGIBILITY:
Inclusion Criteria:

* Mothers must have consented for cord blood collection at delivery
* cord blood must be available for extraction of stem cells.
* >34 weeks gestation
* cord or neonatal pH<7.0 or base deficit>16 milliequivalents per liter (mEq/L) or history of acute perinatal event
* either a 10 minute Apgar < 5 or continued need for ventilation.
* All infants must have signs of encephalopathy within 6 hours of age.

Exclusion Criteria:

* Inability to enroll by 14 days of age.
* Presence of known chromosomal anomaly.
* Presence of major congenital anomalies.
* Severe intrauterine growth restriction (weight <1800g)
* Infants in extremis for whom no additional intensive therapy will be offered by attending neonatologist.
* Parents refuse consent.
* Attending neonatologist refuses consent.
* Failure to collect the infant's cord blood and/or laboratory unable to process cord blood.

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2008-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Adverse event rates occurring in the pilot study population will be compared between the cord blood cell recipients and historical controls. | during infusions: first 18 postnatal days

SECONDARY OUTCOMES:
Secondary endpoints of this pilot study will include preliminary efficacy as measured by neurodevelopmental function at 4 - 6 months and 9 - 12 months of age | 1 year
neuroimaging results will be collected and compared with available results from prior trials of therapies in this population, and from a previously collected set of images from normal term newborns through the first year of life. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Cotten, MD MHS, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Martin PL, Carter SL, Kernan NA, Sahdev I, Wall D, Pietryga D, Wagner JE, Kurtzberg J. Results of the cord blood transplantation study (COBLT): outcomes of unrelated donor umbilical cord blood transplantation in pediatric patients with lysosomal and peroxisomal storage diseases. Biol Blood Marrow Transplant. 2006 Feb;12(2):184-94. doi: 10.1016/j.bbmt.2005.09.016. PMID 16443516
- [Background] Kurtzberg J, Lyerly AD, Sugarman J. Untying the Gordian knot: policies, practices, and ethical issues related to banking of umbilical cord blood. J Clin Invest. 2005 Oct;115(10):2592-7. doi: 10.1172/JCI26690. PMID 16200191
- [Background] Escolar ML, Poe MD, Provenzale JM, Richards KC, Allison J, Wood S, Wenger DA, Pietryga D, Wall D, Champagne M, Morse R, Krivit W, Kurtzberg J. Transplantation of umbilical-cord blood in babies with infantile Krabbe's disease. N Engl J Med. 2005 May 19;352(20):2069-81. doi: 10.1056/NEJMoa042604. PMID 15901860
- [Background] Staba SL, Escolar ML, Poe M, Kim Y, Martin PL, Szabolcs P, Allison-Thacker J, Wood S, Wenger DA, Rubinstein P, Hopwood JJ, Krivit W, Kurtzberg J. Cord-blood transplants from unrelated donors in patients with Hurler's syndrome. N Engl J Med. 2004 May 6;350(19):1960-9. doi: 10.1056/NEJMoa032613. PMID 15128896
- [Background] McGraw P, Liang L, Escolar M, Mukundan S, Kurtzberg J, Provenzale JM. Krabbe disease treated with hematopoietic stem cell transplantation: serial assessment of anisotropy measurements--initial experience. Radiology. 2005 Jul;236(1):221-30. doi: 10.1148/radiol.2353040716. PMID 15987975
- [Result] Cotten CM, Murtha AP, Goldberg RN, Grotegut CA, Smith PB, Goldstein RF, Fisher KA, Gustafson KE, Waters-Pick B, Swamy GK, Rattray B, Tan S, Kurtzberg J. Feasibility of autologous cord blood cells for infants with hypoxic-ischemic encephalopathy. J Pediatr. 2014 May;164(5):973-979.e1. doi: 10.1016/j.jpeds.2013.11.036. Epub 2013 Dec 31. PMID 24388332
- See also: Carolinas Cord Blood Bank web page — http://www.cancer.duke.edu/ccbb/